CLINICAL TRIAL: NCT05484674
Title: Local Control of Hidradenitis Suppurativa After Combination Deroofing and Long-Pulsed 1064-nm Nd:YAG Laser
Brief Title: Control of Hidradenitis Suppurativa of the Underarms After Combination Deroofing and Laser
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000679
Record Dates: First submitted 2022-07-06; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Lasers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One axilla will be treated with deroofing surgery and laser (Experimental): One axilla will be randomly selected for treatment with deroofing surgery and laser while the other axilla will serve as a control with no treatment for each participant
  Interventions: Procedure: Deroofing and laser

INTERVENTIONS:
Procedure: Deroofing and laser — Deroofing and laser to axilla

SUMMARY:
The purpose of the study is to determine whether a series of laser hair removal treatments can improve participant outcomes after deroofing procedures. A deroofing procedure is a surgery where larger hidradenitis suppurativa bumps (called nodules) and hidradenitis suppurativa tunnels (called sinus tracts) are removed and left to heal open without stitches.

DETAILED DESCRIPTION:
Hidradenitis Suppurativa (HS) is a chronic inflammatory disorder characterized by follicular occlusion and rupture which leads to scar and sinus tract formation. Given that medical treatments for HS primarily target inflammation, a multifaceted approach to therapy incorporating procedural techniques is thought to lead to better disease control. Deroofing of nodules and sinus tracts has shown to be beneficial in the treatment of recalcitrant areas that do not respond fully to medical therapy alone. In addition, multiple studies demonstrate the efficacy of long-pulsed 1064-nm Nd:YAG laser in the treatment of HS. To date, no study has evaluated the efficacy of combining surgical deroofing and laser treatment.

In this study, participants with Hurley stage II disease of bilateral axillae who meet the study criteria will be treated. Deroofing will be performed to all nodules and sinus tracts in a randomly selected axilla of each participant. Immediately prior to deroofing, participants will have their initial Nd:YAG laser treatment to the selected axilla. Participants will then be treated every four weeks with a series of additional laser treatments. The opposite (untreated) axilla will serve as a control for monitoring baseline disease activity.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosis of hidradenitis suppurativa Hurley stage II with bilateral axillary involvement
* Must be under the care of a board certified dermatologist and planning to undergo a deroofing procedure of one axilla for the treatment of their HS
* Disease must be active in the bilateral axillae

  * Activity to be defined as having had at least one flare in the last six months
  * Flare to be defined as patient reported worsening of disease beyond baseline or clinical evidence of active inflammation (i.e. erythema, edema, drainage, tenderness)

Exclusion Criteria:

* Pregnancy
* Clinical evidence of active superinfection
* Previous deroofing surgery in any axilla
* Previous laser therapy in any axilla
* Patients on the following medical therapies:

  * Any systemic immunomodulating agent that has been started within 3 months of initial deroofing and laser treatment

    * Patients on immunomodulators >3 months with no change in therapy are eligible for participation
  * Use of topical antibiotics, antiseptics, oral antibiotics, oral steroids, intralesional steroids

    * Patients must have stopped all of these agents at least 2 weeks prior to surgical deroofing
  * Use of intramuscular steroids

    * It must be at least 4 weeks since administration of intramuscular steroids before deroofing for a patient to be eligible for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2022-08-06 (Estimated); Primary Completion 2023-08-06 (Estimated); Study Completion 2023-12-06 (Estimated)

PRIMARY OUTCOMES:
Disease Activity Changes as Assessed by the Hidradenitis Suppurativa Clinical Response | 12 months
  The Hidradenitis Suppurativa Clinical Response (HiSCR) is a validated score defined as a 50% or greater reduction in abscesses and inflammatory nodule counts with no increase in abscesses and draining sinus tracts at the end of the study period, as compared to baseline. A participant will be considered either positive, or achieving HiSCR, which indicates that the study intervention significantly improved the participant's disease, or the patient will be negative, or did not achieve HiSCR, indicating that the intervention did not significantly impact the participant's disease. Study researchers will calculate this score based on clinical assessment and lesion counts assessed at the first study visit and the last two study visits. The percent of participants who achieve HiSCR at the last two study visits will be reported.
Disease Activity Changes as Assessed by the International Hidradenitis Suppurativa Severity Score System | 12 months
  International Hidradenitis Suppurativa Severity Score System (IHS4) changes over the study period will be reported. At each study visit the number of nodules, abscesses, and draining tunnels will be counted in each axilla. The IHS4 score is the number of nodules + abscess count (multiplied by 2) + number of draining tunnels (multiplied by 4). The score can range from 0 lesions and the maximum value is dependent on how many lesions the participant has. The score is used to assess disease severity and can be used to assess how disease severity changes after an intervention. A higher score indicates more active or severe disease, while a lower score indicates less active or less severe disease. Scores throughout the study visits will be reported as well as how these scores change.
Disease Recurrence after the Intervention as Assessed by Clinical Exam | 12 months
  During study visits, a study team member will count the number of nodules, abscesses, and tunnels in each axilla. A higher count indicates more active or severe disease, whereas a lower count indicates less active or less severe disease. Scores can range from 0 lesions to as many as the participant has. Differences between the counts throughout the study visits will be reported.

SECONDARY OUTCOMES:
Quality of Life Changes as Assessed by the Dermatology Quality of Life Index | 12 months
  The Dermatology Life Quality Index (DLQI) tool is a validated questionnaire with 10 questions which asks questions related to activities of daily living and how challenging these are in relation a person's skin disease. Answer choices are either yes or no answers or ratings from "not relevant" or "not at all" to "very much" for each question, regarding how their activities of daily living are affected. Scores range from a minimum of 0 to a maximum of 30 with a higher score indicating a worse quality of life. DLQI surveys will be obtained at the first study visit and the final study visit. Score differences between these two visits will be reported.
Pain as assessed by the Visual Analog Scale | 12 months
  The Visual Analog Scale is a 10-point validated pain scale which allows a patient to choose a score between 0 to 10 with depictions of faces showing emotions, with 0 being no pain and 10 being the worst possible pain. This questionnaire will be administered at various points throughout the study and changes over time will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Venessa Pena-Robichaux, MD, Principal Investigator — Ascension Seton; Courtney Haller, MD, Study Director — University of Texas at Austin

IPD SHARING:
Plan to Share IPD: No